CLINICAL TRIAL: NCT05941975
Title: Multimodal Exploration of Patients With Multiple Sclerosis for an Early Detection of Subtle Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bernard Dachy, Head of neurology department, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-PIRA
Record Dates: First submitted 2023-05-15; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIRA (Experimental): From the MS functional outcome database, identification of a cohort of patients with RMS experiencing progression independent of relapse (PIRA)
  Interventions: Device: Visual Evoked Potential (VEP); Device: Somatosensory evoked potential (SSEP); Device: Transcranial magnetic motor evoked potentials (TCmMEP); Device: Tesla Brain MRI; Diagnostic Test: Blood test - Neurofilament light chain (NfL); Diagnostic Test: Blood test - EBV serology
- N-PIRA (Active Comparator): From the MS functional outcome database, identification of a cohort of patients with RMS not experiencing progression independent of relapse (N-PIRA)
  Interventions: Device: Visual Evoked Potential (VEP); Device: Somatosensory evoked potential (SSEP); Device: Transcranial magnetic motor evoked potentials (TCmMEP); Device: Tesla Brain MRI; Diagnostic Test: Blood test - Neurofilament light chain (NfL); Diagnostic Test: Blood test - EBV serology

INTERVENTIONS:
Device: Visual Evoked Potential (VEP) — To assess the integrity of visual pathways through the optic nerves to the visual cortex, latencies and amplitudes of P100 will be measured after pattern-reversal stimuli.
Device: Somatosensory evoked potential (SSEP) — To assess the integrity of sensitive pathways through the peripheral nerves and dorsal spinal cord to the somatosensory cortex. For the upper limbs, latencies and amplitudes of N9, N13, P14, N20 and P25 will be measured after median nerve stimulation. For the lower limbs, latency and amplitude of P40 will be measured after tibial nerve stimulation.
Device: Transcranial magnetic motor evoked potentials (TCmMEP) — To measure the integrity of motor pathways, the central conduction times will be measured for upper and lower limbs through magnetic stimulations of the primary motor cortex and the spinal cord, at cervical and lumbar levels.
Device: Tesla Brain MRI — All patients will undergo a single brain MRI on a 3T scanner. The acquisition protocol will include high-resolution three-dimensional (3D) T2*-weighted echo-planar imaging and 3D T2-FLAIR images acquired, respectively, during or after intravenous injection of a single dose (0.1mmol/kg) of gadolinium-based contrast material.
Diagnostic Test: Blood test - Neurofilament light chain (NfL) — - Neurofilament light chain (NfL) will be tested (Quanterix's Simoa® Technology) in the serum of patients. To evaluate their variation over time, 3 time-point tests will be obtained at 6 months apart (at baseline, at 6- and 12-month follow-up).
Diagnostic Test: Blood test - EBV serology — EBV serology will be assessed (VCA IgG) in the serum of patients to evaluate the variation of antibody titers over time (at baseline, at 6- and 12-month follow-up), and compare to titers at the time of diagnosis (when available in their medical record).

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory and degenerative disease of the central nervous system (CNS), characterized by a complex interplay of inflammatory demyelination and neuronal damage. The core MS phenotypes defined by clinical course are the relapsing and the progressive forms.Relapsing MS (RMS) is characterized by attacks - also called relapses - defined as new or increasing neurologic dysfunction, followed by periods of partial or complete recovery, without apparent progression of the disease during the periods of remission. In contrast, progressive MS (PMS) is characterized by progressive worsening of neurologic function leading to accumulation of disability over time independent of relapses. Additional descriptors ("active/not-active") serve to better characterize the presence of clinical and/or radiological activity both in relapsing and progressive forms.

In recent years, the concept of a silent progression, also known as smouldering MS, is making its way into the common lexicon of MS experts, challenging the current definitions of MS phenotypes. A growing body of literature suggests that the line between RMS and PMS is not as marked as men thought, and that inflammation and neurodegeneration can represent a single disease continuum coexisting early on in the disease course. Whilst it is established that relapse-associated worsening (RAW) can be accounted for by an acute inflammatory focal damage leading to axonal transection and conduction block, the physiopathology underlying the progression independent of relapse activity (PIRA) remains unclear.

It is becoming apparent that there is an increasing need for a personalized therapeutic approach by considering the individual MS phenotype of each patient, thereby enabling the choice of the molecule best suited to counteract the predominant disease pattern of that individual patient.

There is a limited number of studies combining clinical scores, neurophysiological evaluation and neuroimaging in patients with MS experiencing PIRA. Integrating a multimodal exploration of these patients might allow a step forward in the early recognition, management, and treatment of disability accumulation independent from relapses in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18-year-old with diagnosis of RMS according to 2017 McDonald diagnostic criteria
2. Availability in the functional outcome database of at least 3 time-point complete evaluations with a time frame from the first to the last evaluation of minimum 12 months
3. Most recent functional outcome evaluation within 12 months of enrollment
4. Availability of follow-up MRI data during the observational period

Exclusion Criteria:

a) Contraindication to one or more of the paraclinical tests of the prospective multimodal evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Evoked Potential (VEP) | Change from baseline to 12 months
  To assess the integrity of visual pathways through the optic nerves to the visual cortex.
Somatosensory evoked potential (SSEP) | Change from baseline to 12 months
  To assess the integrity of sensitive pathways through the peripheral nerves and dorsal spinal cord to the somatosensory cortex.
Transcranial magnetic motor evoked potentials (TCmMEP) | Change from baseline to 12 months
  To measure the integrity of motor pathways.
Tesla Brain MRI | Baseline
  Tesla Brain MRI (descriptive outcome)
Neurofilament light chain (NfL) serum levels | Baseline
  Neurofilament light chain (NfL) serum levels
Neurofilament light chain (NfL) serum levels | 6 months after baseline
  Neurofilament light chain (NfL) serum levels
Neurofilament light chain (NfL) serum levels | 12 months after baseline
  Neurofilament light chain (NfL) serum levels
Epstein-Barr virus (EBV) serology (VCA IgG) | Baseline
  EBV serology will be assessed (VCA IgG) in the serum of patients to evaluate the variation of antibody titers over time (at baseline, at 6- and 12-month follow-up), and compare to titers at the time of diagnosis (when available in their medical record).
Epstein-Barr virus (EBV) serology (VCA IgG) | 6 months after baseline
  EBV serology will be assessed (VCA IgG) in the serum of patients to evaluate the variation of antibody titers over time (at baseline, at 6- and 12-month follow-up), and compare to titers at the time of diagnosis (when available in their medical record).
Epstein-Barr virus (EBV) serology (VCA IgG) | 12 months after baseline
  EBV serology will be assessed (VCA IgG) in the serum of patients to evaluate the variation of antibody titers over time (at baseline, at 6- and 12-month follow-up), and compare to titers at the time of diagnosis (when available in their medical record).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No